CLINICAL TRIAL: NCT06186245
Title: Starvation in the Treatment of Diabetic Ketoacidosis: Is There Enough Evidence to Support This Practice?
Brief Title: Starvation in the Treatment of Diabetic Ketoacidosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TTUHSCDKA
Record Dates: First submitted 2023-11-14; First posted 2023-12-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Ketoacidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early feeding (Experimental): If randomized to the experimental group, patient's diet will be advanced to clear liquid for the first day. On the second day, diet will be advanced to full liquid and advanced up to oral (carb controlled 1600 calories) diet as tolerated.
  Interventions: Other: Early feeding with an oral diet
- Nothing per mouth (No Intervention): Patient will be kept without PO intake until they are bridged from the insulin drip

INTERVENTIONS:
Other: Early feeding with an oral diet — Participants in the treatment arm will be initiated on a clear liquid diet on day 1 of medical ICU admission. Diet will be progressed on day 2 to full liquid diet or diabetic diet as patient tolerates based on which diet the patient would prefer.
  Arms: Early feeding

SUMMARY:
Diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state (HHS) are common, but serious metabolic disorders are often encountered in intensive care. In the intensive care setting, it is common to withhold food from patients during treatment of DKA. However, there is no evidence or current literature supporting this practice. The following proposed research investigates the initiation of an early diet versus withholding food during the treatment of diabetic ketoacidosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with the diagnosis of diabetic ketoacidosis (defined as blood glucose greater than 250 mg/dL, arterial pH less than 7.3, serum bicarbonate less than 15 mEq/L, and the presence of ketonemia or ketonuria)
* Age between 18-89
* Admission to the Medical Intensive Care Unit
* Able to provide informed consent

Exclusion Criteria:

* Pregnant and breast-feeding women
* Institutionalized patients or prisoners
* Patients unable to eat by mouth, including intubation, presence of any tube used for enteral feeding (nasogastric tube, orogastric tube, PEG tube, etc.), medical conditions requiring parenteral feeding, and a history of a medical condition that prevented oral intake prior to admission, including achalasia, esophageal cancer, stroke with residual deficits preventing oral intake, amyotrophic lateral sclerosis, or head and neck trauma.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of DKA | Typically resolution of DKA is 24-72 hours, may be up to 5 days in some patients
  Defined as a closed anion gap. Adjusted Anion Gap defined as (Blood Sodium - Blood Chloride - Blood Bicarbonate) + 0.25 x ((normal albumin (4.0)) x (observed albumin)); Elevated Anion Gap is >12
Length of stay in the medical intensive care unit (in days). | Days (Typically 3-5 days in the MICU, may be up to 1 week).
  The time from admission order is placed to the time the transfer to another unit order is placed

SECONDARY OUTCOMES:
Length of stay in the hospital | 3-7 days, may be up to 1-2 weeks.
  from admission order time to the discharge order time
mortality | 30 day
  If patient passes away within 30 days of participating in the study

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kenneth, MD, Principal Investigator — Texas Tech University Health Science Center
Locations (1):
- University Medical Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT06186245/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT06186245/ICF_001.pdf